CLINICAL TRIAL: NCT00425373
Title: A Multi-center, Randomized, Double-blind, Parallel-group, Placebo-controlled, Factorial Study to Evaluate the Efficacy and Safety of 8-week Treatment With Valsartan (40 and 80 mg) and Amlodipine (2.5 and 5 mg) Combined and Alone in Essential Hypertensive Patients
Brief Title: Efficacy and Safety of Valsartan and Amlodipine in Patients With Essential Hypertension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Study Director, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAA489A1301
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Results first posted 2011-02-04 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Essential Hypertension
Keywords: Hypertension, Valsartan, Amlodipine, high blood pressure
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Valsartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (9):
- Valsartan + amlodipine 40/2.5 mg (Experimental)
  Interventions: Drug: Valsartan + amlodipine 40/2.5 mg
- Valsartan + amlodipine 40/5 mg (Experimental)
  Interventions: Drug: Valsartan + amlodipine 40/5 mg
- Valsartan + amlodipine 80/2.5 mg (Experimental)
  Interventions: Drug: Valsartan + amlodipine 80/2.5 mg
- Valsartan + amlodipine 80/5 mg (Experimental)
  Interventions: Drug: Valsartan + amlodipine 80/5 mg
- Valsartan 40 mg (Active Comparator)
  Interventions: Drug: Valsartan 40 mg
- Valsartan 80 mg (Active Comparator)
  Interventions: Drug: Valsartan 80 mg
- Amlodipine 2.5 mg (Active Comparator)
  Interventions: Drug: Amlodipine 2.5 mg
- Amlodipine 5 mg (Active Comparator)
  Interventions: Drug: Amlodipine 5 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valsartan + amlodipine 40/2.5 mg — Valsartan + amlodipine 40/2.5 mg tablet plus 3 tablet and 2 capsule placebos taken once daily
  Arms: Valsartan + amlodipine 40/2.5 mg
Drug: Valsartan + amlodipine 40/5 mg — Valsartan + amlodipine 40/5mg tablet plus 3 tablet and 2 capsule placebos taken once daily
  Arms: Valsartan + amlodipine 40/5 mg
Drug: Valsartan + amlodipine 80/2.5 mg — Valsartan + amlodipine 80/2.5 mg tablet plus 3 tablet and 2 capsule placebos taken once daily
  Arms: Valsartan + amlodipine 80/2.5 mg
Drug: Valsartan + amlodipine 80/5 mg — Valsartan + amlodipine 80/5mg tablet plus 3 tablet and 2 capsule placebos taken once daily
  Arms: Valsartan + amlodipine 80/5 mg
Drug: Valsartan 40 mg — Valsartan 40 mg tablet plus 3 tablet and 2 capsule placebos taken once daily
  Arms: Valsartan 40 mg
Drug: Valsartan 80 mg — Valsartan 80 mg tablet plus 3 tablet and 2 capsule placebos taken once daily
  Arms: Valsartan 80 mg
Drug: Amlodipine 2.5 mg — Amlodipine 2.5 mg capsule plus 4 tablet and 1 capsule placebos taken once daily
  Arms: Amlodipine 2.5 mg
Drug: Amlodipine 5 mg — Amlodipine 5 mg capsule plus 4 tablet and 1 capsule placebos taken once daily
  Arms: Amlodipine 5 mg
Drug: Placebo — 4 tablet and 2 capsule placebos taken once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of fixed combination of valsartan (40 mg and 80 mg) and amlodipine (2.5 mg and 5 mg), valsartan and amlodipine alone, and placebo in reducing blood pressure. The study will investigate the dose response relationship for the combinations, monotherapies, and placebo.

ELIGIBILITY:
Inclusion criteria

* Patients with essential hypertension measured by electronic hemodynamometer. - - Patients must satisfy the following criteria.

  1. MSDBP <110 mmHg and MSSBP <180 mmHg at Visit 1
  2. MSDBP ≥ 90 mmHg and < 110 mmHg and MSSBP < 180 mmHg at Visit 2
  3. MSDBP ≥ 95 mmHg and < 110 mmHg and MSSBP < 180 mmHg at Visit 3
  4. The absolute difference in MSDBP between Visit 2 and 3 is ≤ 10 mmHg
* Male or female outpatients.
* Aged => 20 and =< 80 years (at the time of signing informed consent).
* Patients who have written informed consent to participate in this study.

Exclusion criteria

* Pregnant women, nursing (lactating) mothers, women suspected of being pregnant, or women who wish to be pregnant during the study, women of child-bearing potential.
* Patients with secondary hypertension or suspected of having secondary hypertension.
* Patients with a history of malignant hypertension.
* Patients with an inability to completely discontinue all prior antihypertensive medications safely for a period of 12 weeks as required by the protocol.
* Patients with or with a history of any of the following diseases or signs: Cardiac disease, renal disease, cerebrovascular disorder
* Patients with a clinically significant allergy (asthma on pharmacotherapy, multi-drug allergy, or drug-induced or food-induced anaphylactic reactions).
* Patients hypersensitive to AII receptor antagonists, calcium channel blockers or dihydropyridine derivatives.
* Known moderate or malignant retinopathy.
* Patients with or with a history of pancreatitis. Patients with pancreatic injury, or evidence of impaired pancreatic function/injury within 12 months of Visit 1.
* Patients with any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of any drug.
* Patients with volume depletion based on the investigator's or subinvestigator's clinical judgment using vital signs, skin turgor, moistness of mucous membrane and laboratory values.
* Patients who are found to have low Na and K (Na <130 mEq/L, K <3.3mEq/L) or high in these parameters (Na ≥ 152 mEq/L, K ≥ 5.2 mEq/L) by laboratory tests at Visit 1.
* Patients with type I diabetes mellitus on treatment with insulin, or patients with type II diabetes with poor glucose control defined as a glycosylated hemoglobin (HbA1c) > 8.0% at Visit 1.
* Patients with or with a history of malignant tumors including leukemia and lymphoma, treated or untreated, within the past 5 years of Visit 1 whether or not there is evidence of local recurrence or metastases (except for localized basal cell carcinoma of the skin).
* Patients with any severe, life-threatening disease within the past 5 years. Patients with a history of autoimmune diseases such as rheumatoid arthritis and systemic lupus erythematosus.
* Any surgical or medical condition, which in the opinion of the investigator or subinvestigator, place the patient at higher risk from his/her participation in the study, or are likely to prevent the patient from complying with the requirement of the study or completing the trial period.
* Patients who have with or with a history of drug or alcohol abuse within the last 2 years of Visit 1. Patients who have received other investigational product within 12 weeks of Visit 1.
* Any chronic inflammatory condition needing chronic anti-inflammatory drug therapy.
* Persons directly involved in the execution of this study.
* Patients who are considered unlikely to comply with the requirements specified in the protocol by the investigator or subinvestigator.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1474 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Japan, Study Chair — Sponsor GmbH
Locations (1):
- Novartis Pharmaceuticals, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valsartan + Amlodipine 40/2.5 mg | Valsartan + Amlodipine 40/5 mg | Valsartan + Amlodipine 80/2.5 mg | Valsartan + Amlodipine 80/5 mg | Valsartan 40 mg | Valsartan 80 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Placebo
Started | 159 | 167 | 160 | 162 | 169 | 163 | 161 | 161 | 166
Completed | 154 | 164 | 157 | 160 | 159 | 154 | 154 | 151 | 148
Not Completed | 5 | 3 | 3 | 2 | 10 | 9 | 7 | 10 | 18
Not completed — Adverse Event | 2 | 2 | 0 | 1 | 4 | 6 | 2 | 3 | 8
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 1 | 4 | 0 | 2 | 2 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan + Amlodipine 40/2.5 mg | Valsartan + Amlodipine 40/5 mg | Valsartan + Amlodipine 80/2.5 mg | Valsartan + Amlodipine 80/5 mg | Valsartan 40 mg | Valsartan 80 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Placebo | Total
Number analyzed (Participants) | 159 | 167 | 160 | 162 | 169 | 163 | 161 | 161 | 166 | 1468
Age Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.34) | 52.8 (10.70) | 52.8 (10.76) | 54.1 (9.75) | 52.9 (10.08) | 52.6 (11.29) | 53.2 (10.83) | 54.4 (10.67) | 51.5 (10.58) | 53.1 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 49 | 40 | 39 | 38 | 49 | 49 | 40 | 55 | 405
  Male | 113 | 118 | 120 | 123 | 131 | 114 | 112 | 121 | 111 | 1063

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (MSDBP) From Baseline to End of Study (Week 8)
Description: At study entry, blood pressure was measured in both arms using a standard method described in the protocol. The arm with the higher diastolic BP reading was used for the measurements at all subsequent visits. Blood pressure in the sitting position was measured after resting in a seated position for at least 5 minutes. The measurement was repeated a total of 3 times at intervals of 1 to 2 minutes. A negative number indicates lowered blood pressure.
Time Frame: Baseline to end of study (Week 8)
Population: Intent-to-treat (ITT): All randomized patients who had a baseline and at least one post-baseline assessment of the variable analyzed. Baseline is the Week 0 value and end of study is the value at Week 8 or the last observation carried forward (LOCF) value.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Valsartan + Amlodipine 40/2.5 mg | Valsartan + Amlodipine 40/5 mg | Valsartan + Amlodipine 80/2.5 mg | Valsartan + Amlodipine 80/5 mg | Valsartan 40 mg | Valsartan 80 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Placebo
Number analyzed (Participants) | 159 | 167 | 160 | 162 | 169 | 163 | 161 | 161 | 166
mm Hg | -13.5 (0.62) | -16.5 (0.60) | -12.6 (0.62) | -17.0 (0.61) | -8.5 (0.60) | -8.8 (0.61) | -10.3 (0.61) | -13.4 (0.61) | -4.8 (0.61)

2. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (MSSBP) From Baseline to End of Study (Week 8)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Valsartan + Amlodipine 40/2.5 mg | Valsartan + Amlodipine 40/5 mg | Valsartan + Amlodipine 80/2.5 mg | Valsartan + Amlodipine 80/5 mg | Valsartan 40 mg | Valsartan 80 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Placebo
Number analyzed (Participants) | 159 | 167 | 160 | 162 | 169 | 163 | 161 | 161 | 166
mm Hg | -16.7 (0.88) | -22.0 (0.86) | -16.9 (0.88) | -22.9 (0.87) | -9.3 (0.85) | -9.5 (0.87) | -13.6 (0.87) | -16.6 (0.87) | -4.4 (0.86)

3. Secondary Outcome: Percentage of Patients Achieving MSDBP < 90 mmHg or a => 10 mm Hg Decrease Compared to Baseline at the End of the Study (Week 8)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan + Amlodipine 40/2.5 mg | Valsartan + Amlodipine 40/5 mg | Valsartan + Amlodipine 80/2.5 mg | Valsartan + Amlodipine 80/5 mg | Valsartan 40 mg | Valsartan 80 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Placebo
Number analyzed (Participants) | 159 | 167 | 160 | 162 | 169 | 163 | 161 | 161 | 166
Percentage of patients | 77.4 | 88.0 | 80.6 | 86.4 | 52.1 | 47.9 | 62.1 | 74.5 | 36.1

4. Secondary Outcome: Percentage of Patients Achieving MSDBP < 90mmHg at the End of the Study (Week 8)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan + Amlodipine 40/2.5 mg | Valsartan + Amlodipine 40/5 mg | Valsartan + Amlodipine 80/2.5 mg | Valsartan + Amlodipine 80/5 mg | Valsartan 40 mg | Valsartan 80 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Placebo
Number analyzed (Participants) | 159 | 167 | 160 | 162 | 169 | 163 | 161 | 161 | 166
Percentage of patients | 67.3 | 82.6 | 72.5 | 80.9 | 46.2 | 41.1 | 55.3 | 67.1 | 31.9

5. Secondary Outcome: Percentage of Patients Achieving MSDBP < 90 mm Hg and MSSBP < 140 mm Hg at the End of the Study (Week 8)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan + Amlodipine 40/2.5 mg | Valsartan + Amlodipine 40/5 mg | Valsartan + Amlodipine 80/2.5 mg | Valsartan + Amlodipine 80/5 mg | Valsartan 40 mg | Valsartan 80 mg | Amlodipine 2.5 mg | Amlodipine 5 mg | Placebo
Number analyzed (Participants) | 159 | 167 | 160 | 162 | 169 | 163 | 161 | 161 | 166
Percentage of patients | 55.3 | 75.4 | 59.4 | 72.2 | 33.1 | 30.1 | 41.0 | 57.1 | 18.7

ADVERSE EVENTS:
Groups:
- Amlodipine 5 mg: Amlodipine 2.5 mg 2 capsules plus 4 tablet placebos taken once daily
Arm/Group | Placebo | Valsartan 40 mg | Valsartan 80 mg | Amlodipine 2.5 mg | Valsartan + Amlodipine 40/2.5 mg | Valsartan + Amlodipine 80/2.5 mg | Amlodipine 5 mg | Valsartan + Amlodipine 40/5 mg | Valsartan + Amlodipine 80/5 mg
Serious Adverse Events (participants affected / at risk) | 2/166 | 0/169 | 0/163 | 1/161 | 0/159 | 1/160 | 0/161 | 1/167 | 0/162
Other Adverse Events (participants affected / at risk) | 17/166 | 23/169 | 19/163 | 12/161 | 17/159 | 9/160 | 12/161 | 20/167 | 14/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=166) | Valsartan 40 mg (N=169) | Valsartan 80 mg (N=163) | Amlodipine 2.5 mg (N=161) | Valsartan + Amlodipine 40/2.5 mg (N=159) | Valsartan + Amlodipine 80/2.5 mg (N=160) | Amlodipine 5 mg (N=161) | Valsartan + Amlodipine 40/5 mg (N=167) | Valsartan + Amlodipine 80/5 mg (N=162)
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=166) | Valsartan 40 mg (N=169) | Valsartan 80 mg (N=163) | Amlodipine 2.5 mg (N=161) | Valsartan + Amlodipine 40/2.5 mg (N=159) | Valsartan + Amlodipine 80/2.5 mg (N=160) | Amlodipine 5 mg (N=161) | Valsartan + Amlodipine 40/5 mg (N=167) | Valsartan + Amlodipine 80/5 mg (N=162)
Nasopharyngitis (Infections and infestations) | 17 | 23 | 19 | 12 | 17 | 9 | 12 | 20 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.